CLINICAL TRIAL: NCT05895643
Title: Does the Glucagon-like Peptide 1 (GLP-1) Receptor Agonist Semaglutide Reduce Alcohol Intake in Patients With Alcohol Use Disorder and Comorbid Obesity?
Brief Title: Does Semaglutide Reduce Alcohol Intake in Patients With Alcohol Use Disorder and Comorbid Obesity?
Acronym: SEMALCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Psychiatric Centre Rigshospitalet (Other)
Collaborators: Neurobiology Research Unit (Unknown)
Responsible Party: Principal Investigator, Anders Fink-Jensen, MD, DMSci, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: The SEMALCO study; U1111-1286-6919 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2023-05-26; First posted 2023-06-08 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Abuse; Alcohol Addiction; Alcohol Dependence; Alcohol Use Disorder
Keywords: GLP-1; Glucagon-like peptide 1; semaglutide; fMRI; MRS
MeSH Terms: conditions — Alcoholism | interventions — semaglutide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- semaglutide (Experimental): Wegovy once-weekly s.c.titrated to a maximum dose of 2.4 mg
  Interventions: Drug: Semaglutide Injectable Product
- placebo (Placebo Comparator): Saline s.c. once-weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Injectable Product — Once weekly injections s.c with semaglutide (Wegovy)
  Other Names: Wegovy
  Arms: semaglutide
Drug: Placebo — Once weekly injections s.c with placebo (BD Posiflush)
  Other Names: BD Posiflush (saline)
  Arms: placebo

SUMMARY:
This 26-week long, double-blinded randomized clinical trial aims to investigate the effects of the GLP-1 receptor agonist semaglutide s.c. vs placebo on alcohol consumption in 108 patients diagnosed with alcohol use disorder and comorbid obesity (BMI>30 kg/m2).

Patients will be treated for 26 weeks with semaglutide subcutaneously (s.c.) once weekly or placebo. The medication will be provided as a supplement to standardised cognitive behavioural therapy. A subgroup of the patients will have two brain scans (Magnetic Resonance Spectroscopy (MRS) and functional Magnetic Resonance Imaging (fMRI)) conducted in one scan session at week 0 and 26.

The primary endpoint is the percentage-point reduction in total number of heavy drinking days, defined as days with an excess intake of 48/60 grams of alcohol per day (women and men, respectively) from baseline to follow-up after 26 weeks of treatment, measured by the timeline followback (TLFB) method.

ELIGIBILITY:
Inclusion Criteria:

* Informed oral and written consent
* Diagnosed with alcohol dependence according to the criteria of the International Classification of Diseases 10 (ICD-10), and diagnosed with alcohol use disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Alcohol use disorder identification test (AUDIT) score >15
* Body mass index (BMI) above or equal to 30 kg/m2
* Age 18 - 70 years (both included)
* Heavy alcohol drinking defined as more than 6 days with alcohol consumption over 4 units (48 g alcohol) for women and 5 units (60 g alcohol) for men during a consecutive 30-day period, within 40 days prior to baseline evaluation, measured by the TLFB method. The 30-day period will be the 30 consecutive days with the biggest alcohol intake (most heavy drinking days and the largest amount of total alcohol) out of the 40 days.

Exclusion Criteria:

* Severe psychiatric disease, defined as a diagnosis of schizophrenia, paranoid psychosis, bipolar disorder or mental retardation
* A history of delirium tremens or alcohol withdrawal seizures
* No serious withdrawal symptoms at inclusion (a score higher than 9 on the Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar)) at baseline examinations
* Present or former neurological disease, including traumatic brain injury
* Type 1 diabetes, type 2 diabetes in poor glycaemic control (defined as HbA1c ≥48 mmol/l or fasting plasma glucose above 7.0 mmol/l at inclusion)
* Females of childbearing potential who are pregnant, breast-feeding or have the intention of becoming pregnant within the next 9 months (26 weeks plus two months after discontinuation of semaglutide), or are not using contraceptives (during the whole study period) considered as highly effective (combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) intrauterine device, bilateral tubal occlusion, vasectomised partner, sexual abstinence).
* Pregnancy (serum human chorionic gonadotropin (hCG) > 3 U/L at inclusion)
* Impaired hepatic function (liver transaminases >3 times the upper limit)
* Impaired renal function (eGFR < 50 ml/min and/or plasma creatinine >150 μmol/l)
* Impaired pancreatic function (any history of acute or chronic pancreatitis and/or amylase > 2 times upper limit)
* Former medullary thyroid carcinoma (MTC) and/or family history with MTC and/or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
* Cardiac problems defined as decompensated heart failure (NYHA class III or IV), unstable angina pectoris and/or myocardial infarction within the last 12 months
* Uncontrolled hypertension (systolic blood pressure >180 mmHg, diastolic blood pressure >110 mmHg)
* Concomitant pharmacotherapy against alcohol use disorder, i.e., disulfiram, naltrexone, acamprosate, or nalmefene, since the first of the 30 drinking days registered for inclusion at the TLFB-schedule.
* Receiving any investigational drug within the last three months
* Use of weight-lowering pharmacotherapy within the preceding 3 months
* Any other active substance use defined as a DUDIT-score >1 (except nicotine)
* Hypersensitivity to the active substance or any of the excipients
* Only for patients undergoing brain scans:

  o Contraindications for undergoing an MRI scan (magnetic implants, pacemaker, claustrophobia, etc.)
* Unable to speak and/or understand Danish
* Any condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in heavy drinking days | From baseline to 26 weeks of treatment
  Change in alcohol consumption, defined as the change in percentage of heavy drinking days during a period of 30 consecutive days, after 26 weeks of treatment adjusted for baseline (percentage points (pp)). A heavy drinking day is defined as more than 60/48 grams (men/women) of alcohol in one day, measured with the validated timeline follow-back (TLFB) method.

SECONDARY OUTCOMES:
Change in heavy drinking days adjusted for maximum tolerable semaglutide dose given | From baseline to 26 weeks of treatment
  Change in heavy drinking days during a period of 30 consecutive days, after 26 weeks of treatment adjusted for baseline (percentage points (pp)) and maximum tolerable semaglutide dose given.
Change in heavy drinking days adjusted for weightloss | From baseline to 26 weeks of treatment
  Change in heavy drinking days during a period of 30 consecutive days, after 26 weeks of treatment adjusted for baseline (percentage points (pp)) and weight loss during the 26 weeks of treatment
Total alcohol consumption | From baseline to 26 weeks of treatment
  Change in total alcohol consumption /gram/last 30 consecutive days)
Drinks per day | From baseline to 26 weeks of treatment
  Change in total drinks per day (last 30 consecutive days)
Days without alcohol consumption | From baseline to 26 weeks of treatment
  Number of days without alcohol consumption in the last 30 consecutive days
Time to relapse | From baseline to 26 weeks of treatment
  Time to relapse, defined as the time to first alcohol intake
Time to relapse (heavy drinking day) | From baseline to 26 weeks of treatment
  Time to first heavy drinking day
World Health Organization (WHO) Risk Levels of Alcohol Consumption | From baseline to 26 weeks of treatment
  Change in WHO alcohol risk level in the last 30 consecutive days, measured with the validated timeline follow-back (TLFB) method.
Penn Alcohol Craving Scale (PACS) score | From baseline to 26 weeks of treatment
  Change in Penn Alcohol Craving Scale (PACS) score. Minimum score = 0, maximum score =30. A high score means a worse outcome.
Alcohol Use Disorder Identification Test (AUDIT) score | From baseline to 26 weeks of treatment
  Change in Alcohol Use Disorder Identification Test (AUDIT) score. Minimum score = 0, maximum score =40. A high score means a worse outcome.
Drug Use Disorders Identification Test (DUDIT) score | From baseline to 26 weeks of treatment
  Change in Drug Use Disorders Identification Test (DUDIT) score. Minimum score = 0, maximum score =44. A high score means a worse outcome.
Fibrosis-4 (FIB4) score | From baseline to 26 weeks of treatment
  Change in Fibrosis-4 (FIB4) score, calculated from the parameters: the patient's age, blood aspartate aminotransferase levels (ASAT), thrombocytes and alanine transaminase (ALAT). A higher score means a worse outcome.
Measure of life quality - World Health Organization Quality of Life brief (WHOQOL-BREF) score | From baseline to 26 weeks of treatment
  Change in Measures of Health (WHOQOL-BREF) score. Minimum score = 26, maximum score =130. Higher scores mean a better outcome in items 1-2 + 10-25. A higher score in items 3-9 + 26 means a worse outcome.
Fagerströms Test for Nicotine Dependence score | From baseline to 26 weeks of treatment
  Change in Fagerströms Test for Nicotine Dependence score. Minimum score = 0, maximum score =10. A high score means a worse outcome.
Gamma-glutamyl transferase (GGT) | From baseline to 26 weeks of treatment
  Change in blood gamma-glutamyl transferase (GGT)
Alanine transaminase (ALAT) | From baseline to 26 weeks of treatment
  Change in blood alanine transaminase (ALAT)
Phosphatidyl ethanol (PEth) | From baseline to 26 weeks of treatment
  Change in plasma levels of phosphatidyl ethanol (PEth)
Mean cell volume (MCV) | From baseline to 26 weeks of treatment
  Change in blood mean cell volume (MCV)
Body weight | From baseline to 26 weeks of treatment
  Change in Body weight
Blood pressure | From baseline to 26 weeks of treatment
  Change in blood pressure (both systolic and diastolic)
Pulse | From baseline to 26 weeks of treatment
  Change in pulse
Waist circumference | From baseline to 26 weeks of treatment
  Change in waist circumference
Glycaemic control parameters | From baseline to 26 weeks of treatment
  Change in HbA1c
MRS brain gamma-aminobutyric acid (GABA) levels | From baseline to 26 weeks of treatment
  Change in brain GABA levels (cortical, caudate, and putamen) assessed by MRS brain scans
fMRI alcohol cue-reactivity | From baseline to 26 weeks of treatment
  Change in brain alcohol cue-response in reward-processing brain regions (ventral and dorsal striatum, puta-men, nucleus accumbens, and caudate), including the septal area assessed by fMRI brain scans

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fink-Jensen, MD, DMSc, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Psychiatric Center Copenhagen, Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Jensen ME, Klausen MK, Bergmann ML, Knudsen GM, Vilsboll T, Stove C, Fink-Jensen A. Blood phosphatidylethanol measurements indicate GLP-1 receptor stimulation causes delayed decreases in alcohol consumption. Alcohol Clin Exp Res (Hoboken). 2025 May;49(5):1161-1165. doi: 10.1111/acer.70041. Epub 2025 Mar 23. PMID 40123107
- [Derived] Klausen MK, Kuzey T, Pedersen JN, Justesen SK, Rasmussen L, Knorr UB, Mason G, Ekstrom CT, Holst JJ, Koob G, Benveniste H, Volkow ND, Knudsen GM, Vilsboll T, Fink-Jensen A. Does semaglutide reduce alcohol intake in Danish patients with alcohol use disorder and comorbid obesity? Trial protocol of a randomised, double-blinded, placebo-controlled clinical trial (the SEMALCO trial). BMJ Open. 2025 Jan 8;15(1):e086454. doi: 10.1136/bmjopen-2024-086454. PMID 39779270

DOCUMENTS (2):
  • Study Protocol (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT05895643/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT05895643/SAP_002.pdf